CLINICAL TRIAL: NCT00849732
Title: A Worldwide, Phase I, Dose-Escalating Study of Safety, Tolerability, and Immunogenicity of a 3-Dose Regimen of the MRKAd5 HIV-1 Gag Vaccine in Healthy Adults
Brief Title: A Worldwide, Phase I, Dose-Escalating Study of a 3-Dose Regimen of the MRKAd5 (Clade B) Vaccine in Healthy Adults (V520-018)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: HIV Vaccine Trials Network (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V520-018; 2009_549
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: HIV-1; HIV Infections
Keywords: HIV Seronegativity; Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): V520 (1x10^9 vp/d)
  Interventions: Biological: V520; Biological: Comparator: V520 (1x10^9 vp/d)
- 2 (Experimental): V520 (1x10^10 vp/d)
  Interventions: Biological: Comparator: V520 (1x10^10 vp/d)
- 3 (Placebo Comparator): Placebo to V520
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: V520 — Intentionally Blank
  Arms: 1
Biological: Comparator: V520 (1x10^9 vp/d) — 1.0 mL intramuscular injection of MRKAd5 HIV-1 gag vaccine at 1x10^9 vp/d given at Day 1, Week 4, and Week 26
  Arms: 1
Biological: Comparator: V520 (1x10^10 vp/d) — 1.0 mL intramuscular injection of MRKAd5 HIV-1 gag vaccine at 1x10^10 vp/d given at Day 1, Week 4, and Week 26
  Arms: 2
Biological: Comparator: Placebo — Placebo to MRKAd5 HIV-1 gag vaccine 1.0 mL intramuscular injection given at Day 1, Week 4, and Week 26
  Arms: 3

SUMMARY:
This three stage study will evaluate the safety and tolerability of MRKAd5 HIV-1 Gag Vaccine. In Stage I subjects will be randomized to receive the vaccine at 1x10^9 viral particles/dose (vp/d) or placebo. In Stage II subjects will be randomized to receive the vaccine at 1x10^10 vp/d or placebo. In Stage III subjects will be randomized to receive the vaccine at 1x10^9 vp/d, at 1x10^10 vp/d, or placebo. Immunogenicity of the single dose regimen of MRKAd5 HIV-1 Gag Vaccine will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good general health
* Subject tests negative for Hepatitis B, Hepatitis C, and HIV
* Subjects of reproductive potential agree to use an accepted method of birth control through the entire study

Exclusion Criteria:

* Subject has a recent history of fever at time of vaccination
* Subject has received immune globulin or blood product 3 months prior to injection
* Subject has been vaccinated with live virus vaccine 30 days prior to receipt of first dose
* Subject has been vaccinated with inactivated vaccine with 14 days prior to receipt of first dose
* Subject has a chronic medical condition that is considered progressive
* Subject has history of malignancy
* Subject weighs less than 105 lb.
* Female subject is pregnant or breast feeding, Male subject is planning to impregnate during the first year of study
* Subject has contraindication to intramuscular injection
* Subject is unlikely or unwilling to adhere to lower risk sex practices during the course of the study
* Subject has a tattoo on the deltoid region of the arm or the injection of Depo-Provera

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 3 dose prime-boost regimen of MRKAd5 HIV-1 gag vaccine | 4 weeks after third vaccination

SECONDARY OUTCOMES:
breadth of immune response measured by several assays | 4 weeks after third vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Nicholson O, DiCandilo F, Kublin J, Sun X, Quirk E, Miller M, Gray G, Pape J, Robertson MN, Mehrotra DV, Self S, Turner K, Sanchez J, Pitisuttithum P, Duerr A, Dubey S, Kierstead L, Casimiro D, Hammer For The Merck V/Hiv Vaccine Trials Network Study Team SM. Safety and Immunogenicity of the MRKAd5 gag HIV Type 1 Vaccine in a Worldwide Phase 1 Study of Healthy Adults. AIDS Res Hum Retroviruses. 2011 May;27(5):557-567. doi: 10.1089/AID.2010.0151. Epub 2010 Nov 23. PMID 20854108
- [Derived] Pine SO, Kublin JG, Hammer SM, Borgerding J, Huang Y, Casimiro DR, McElrath MJ. Pre-existing adenovirus immunity modifies a complex mixed Th1 and Th2 cytokine response to an Ad5/HIV-1 vaccine candidate in humans. PLoS One. 2011 Apr 13;6(4):e18526. doi: 10.1371/journal.pone.0018526. PMID 21533229